CLINICAL TRIAL: NCT06052267
Title: A Randomized, Double-Blind, Multicenter, Active-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Fluticasone Propionate/Albuterol Sulfate Fixed-Dose Combination on Severe Asthma Exacerbations in Patients With Asthma
Brief Title: A Study to Test if a Fixed-Dose Combination of Fluticasone Propionate/Albuterol Sulfate is Effective in Preventing Asthma Exacerbations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FpA-AS-30094; 2023-505435-12-00 (Other: EUCT)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TEV-56248 Low Dose (Experimental): Inhalation powder via multidose dry powder inhaler with integrated electronic module (eMDPI) with a dosing frequency of 2 inhalations as needed to control asthma symptoms.
  Interventions: Drug: TEV-56248
- TEV-56248 High Dose (Experimental): Inhalation powder via multidose dry powder inhaler with integrated electronic module (eMDPI) with a dosing frequency of 2 inhalations as needed to control asthma symptoms.
  Interventions: Drug: TEV-56248
- Albuterol sulfate (Active Comparator): Inhalation powder via multidose dry powder inhaler with integrated electronic module (eMDPI) with a dosing frequency of 2 inhalations as needed to control asthma symptoms.
  Interventions: Drug: Albuterol sulfate

INTERVENTIONS:
Drug: TEV-56248 — Fluticasone Propionate/Salbutamol Sulfate. Oral inhalation powder.
  Arms: TEV-56248 High Dose; TEV-56248 Low Dose
Drug: Albuterol sulfate — Oral inhalation powder
  Arms: Albuterol sulfate

SUMMARY:
The primary objective of the study is to assess the efficacy of high dose fluticasone propionate (Fp)/albuterol sulfate (ABS) integrated electronic module multidose dry powder inhaler (eMDPI) compared to ABS eMDPI in decreasing severe clinical asthma exacerbation (CAEs).

Secondary Objectives:

To evaluate the efficacy of Fp/ABS low dose compared to ABS and the effect on systemic corticosteroid (SCS) exposure

To evaluate the safety and tolerability of Fp/A BS

The duration for each participant will be a minimum of 28 weeks including 2 weeks of screening, 2-4 weeks of run-in period and a double blind treatment period of minimum 24 weeks, however due to the event-driven nature of this study, the duration may range up to approximately 42 months depending on the timing when the participant was enrolled to the study, and when the study reaches its completion criteria

ELIGIBILITY:
Inclusion Criteria:

* The participant has a documented diagnosis of asthma for at least 1 year according to the 2022 GINA guidelines.
* The participant has a documented history of at least 1 severe clinical asthma exacerbation (CAE) ending within the past 12 month.
* The participant is using any prescribed inhaled asthma controller medication (at a stable dose for 1 month prior to the screening visit).
* If female, the participant is currently not pregnant, breastfeeding, or attempting to become pregnant (for at least 30 days before the screening visit and throughout the duration of the study), or is of nonchildbearing potential

NOTE- Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* The participant has life-threatening asthma defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s) within 5 years before screening.
* The participant has a suspected bacterial or viral infection (other than Coronavirus Disease [COVID-19]) of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the screening period.
* Participants with a confirmed infection with COVID-19 within 6 weeks prior to the screening visit, or with residual COVID-19 symptoms ("long COVID-19").
* The participant has had a clinical asthma exacerbation (CAE) requiring systemic corticosteroids within 30 days before screening, or any hospitalization for asthma within 2 months before screening.
* The participant is a current smoker and/or has a history of ≥10 pack years history of smoking. A current smoker is defined as any participant who has used any form of tobacco product (including oral) within the past 6 months.
* The participant has significantly abused alcohol and/or illicit prohibited drugs within the previous 24 months.
* The participant has participated as a randomized participant in any investigational drug study within 30 days.
* The participant has been hospitalized for psychiatric disorder or attempted suicide within 1 year of screening.

NOTE- Additional criteria apply, please contact the investigator for more information

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Severe Clinical Asthma Exacerbation (CAE) with High Dose (HD) Fp/ABS eMDPI | Up to 42 months

SECONDARY OUTCOMES:
Time to first severe CAE with Low Dose (LD) Fp/ABS eMDPI | Up to 42 months
Annualized Severe CAE Rate | Up to 42 months
  Annualized severe CAE rate is calculated for each participant as the sum of total number of CAE events divided by the duration of follow up time (years).
Total Annualized SCS Exposure Over the Treatment Period | Up to 42 months
  Total annualized SCS exposure will be calculated for each participant as the sum of the cumulative doses of SCS divided by the duration of time (years) the participant was in the treatment period, from randomization and up to end of treatment.
Asthma Control Questionnaire-5 (ACQ-5) Response | Baseline, Week 24
  Response is defined as achieving a decrease in score from baseline value of at least 0.5 (participants aged ≥6 years).
  The ACQ-5 is a shortened version of the validated asthma assessment tool (ie, ACQ) and includes 5 questions that are self-assessments (completed by the participant). Each item on the ACQ-5 has a possible score ranging from 0 to 6, and the total score is the mean of all responses.
Composite Responders Based on Asthma Quality of Life Questionnaire + 12 (AQLQ+12) or Pediatric AQLQ (PAQLQ) | Baseline, Week 24
  Responders are defined as the composite of participants achieving an increase in score from baseline of at least 0.5 on the AQLQ+12 or PAQLQ (participants aged ≥7 years).
  The AQLQ + 12 is a modified version of the standardized AQLQ, which was developed to measure functional impairments experienced by adults ≥17 years of age. The AQLQ + 12 is valid for participants aged 12 to 70 years and includes 32 questions in 4 domains (symptoms, activity limitation, emotional function, and environmental stimuli). Responses are rated on a 7-point scale where 7 = no impairment and 1 = severe impairment.
  The PAQLQ Questionnaire includes 23 items in 3 domains (symptoms, activity limitation, emotional function) and a 7-point scale (7 = not bothered at all; 1 = extremely bothered). It is intended for participants ages 7-11.
Number of Participants with at Least One Adverse Event | Up to 42 months
  Adverse events include clinically significant changes in clinical laboratory test results (serum chemistry, hematology, and urinalysis), vital signs measurements (blood pressure, pulse rate, body temperature, and respiratory rate), and 12-lead electrocardiogram (ECG) findings.
Number of Participants with at Least One Serious Adverse Event | Up to 42 months
Number of Participants Who Withdrew From the Trial Due to Treatment-Emergent Adverse Events | Up to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (393):
- United States (157):
  - Teva Investigational Site 15706, Birmingham, Alabama
  - Teva Investigational Site 15786, Birmingham, Alabama
  - Teva Investigational Site 15768, Dothan, Alabama
  - Teva Investigational Site 15581, Paradise Valley, Arizona
  - Teva Investigational Site 15710, Scottsdale, Arizona
  - Teva Investigational Site 15661, Tucson, Arizona
  - Teva Investigational Site 15685, Bakersfield, California
  - Teva Investigational Site 15721, Fresno, California
  - Teva Investigational Site 15788, Huntington Beach, California
  - Teva Investigational Site 15720, La Jolla, California
  - Teva Investigational Site 15687, La Palma, California
  - Teva Investigational Site 15708, Long Beach, California
  - Teva Investigational Site 15712, Long Beach, California
  - Teva Investigational Site 15643, Los Angeles, California
  - Teva Investigational Site 15695, Napa, California
  - Teva Investigational Site 15692, Northridge, California
  - Teva Investigational Site 15682, Redondo Beach, California
  - Teva Investigational Site 15629, San Bernardino, California
  - Teva Investigational Site 15709, San Diego, California
  - Teva Investigational Site 15704, San Jose, California
  - Teva Investigational Site 15620, Stockton, California
  - Teva Investigational Site 15621, Westminster, California
  - Teva Investigational Site 15612, Aurora, Colorado
  - Teva Investigational Site 15588, Colorado Springs, Colorado
  - Teva Investigational Site 15765, Colorado Springs, Colorado
  - Teva Investigational Site 15676, Englewood, Colorado
  - Teva Investigational Site 15781, Washington D.C., District of Columbia
  - Teva Investigational Site 15660, Aventura, Florida
  - Teva Investigational Site 15624, Cape Coral, Florida
  - Teva Investigational Site 15598, Cutler Bay, Florida
  - Teva Investigational Site 15776, Doral, Florida
  - Teva Investigational Site 15579, Greenacres City, Florida
  - Teva Investigational Site 15582, Hialeah, Florida
  - Teva Investigational Site 15664, Hialeah, Florida
  - Teva Investigational Site 15657, Homestead, Florida
  - Teva Investigational Site 15713, Jacksonville, Florida
  - Teva Investigational Site 15632, Leesburg, Florida
  - Teva Investigational Site 15777, Margate, Florida
  - Teva Investigational Site 15602, Miami, Florida
  - Teva Investigational Site 15722, Miami, Florida
  - Teva Investigational Site 15724, Miami, Florida
  - Teva Investigational Site 15655, Miami, Florida
  - Teva Investigational Site 15605, Miami, Florida
  - Teva Investigational Site 15634, Miami, Florida
  - Teva Investigational Site 15596, Miami, Florida
  - Teva Investigational Site 15654, Miami, Florida
  - Teva Investigational Site 15773, Miami, Florida
  - Teva Investigational Site 15652, Miami, Florida
  - Teva Investigational Site 15585, Miami, Florida
  - Teva Investigational Site 15639, Miami, Florida
  - Teva Investigational Site 15645, Miami, Florida
  - Teva Investigational Site 15772, Miami, Florida
  - Teva Investigational Site 15592, Miami, Florida
  - Teva Investigational Site 15769, Miami, Florida
  - Teva Investigational Site 15644, Miami, Florida
  - Teva Investigational Site 15589, Miami Lakes, Florida
  - Teva Investigational Site 15599, Miami Lakes, Florida
  - Teva Investigational Site 15595, Miami Lakes, Florida
  - Teva Investigational Site 15665, Oldsmar, Florida
  - Teva Investigational Site 15659, Orlando, Florida
  - Teva Investigational Site 15617, Orlando, Florida
  - Teva Investigational Site 15625, Orlando, Florida
  - Teva Investigational Site 15597, Pembroke Pines, Florida
  - Teva Investigational Site 15767, Sweetwater, Florida
  - Teva Investigational Site 15587, Tamarac, Florida
  - Teva Investigational Site 15611, Tampa, Florida
  - Teva Investigational Site 15619, Tampa, Florida
  - Teva Investigational Site 15653, Tampa, Florida
  - Teva Investigational Site 15606, Winter Park, Florida
  - Teva Investigational Site 15717, Atlanta, Georgia
  - Teva Investigational Site 15711, Conyers, Georgia
  - Teva Investigational Site 15626, Savannah, Georgia
  - Teva Investigational Site 15604, Boise, Idaho
  - Teva Investigational Site 15669, Chicago, Illinois
  - Teva Investigational Site 15616, Chicago, Illinois
  - Teva Investigational Site 15716, Chicago, Illinois
  - Teva Investigational Site 15600, Skokie, Illinois
  - Teva Investigational Site 15674, Evansville, Indiana
  - Teva Investigational Site 15580, Overland Park, Kansas
  - Teva Investigational Site 15627, Lexington, Kentucky
  - Teva Investigational Site 15770, Lafayette, Louisiana
  - Teva Investigational Site 15667, Bangor, Maine
  - Teva Investigational Site 15689, Rockville, Maryland
  - Teva Investigational Site 15583, White Marsh, Maryland
  - Teva Investigational Site 15628, Boston, Massachusetts
  - Teva Investigational Site 15686, Fall River, Massachusetts
  - Teva Investigational Site 15663, North Dartmouth, Massachusetts
  - Teva Investigational Site 15764, South Dartmouth, Massachusetts
  - Teva Investigational Site 15702, Detroit, Michigan
  - Teva Investigational Site 15701, Flint, Michigan
  - Teva Investigational Site 15593, Ypsilanti, Michigan
  - Teva Investigational Site 15648, Kansas City, Missouri
  - Teva Investigational Site 15640, St Louis, Missouri
  - Teva Investigational Site 15650, St Louis, Missouri
  - Teva Investigational Site 15633, St Louis, Missouri
  - Teva Investigational Site 15790, Hastings, Nebraska
  - Teva Investigational Site 15679, Las Vegas, Nevada
  - Teva Investigational Site 15725, North Bergen, New Jersey
  - Teva Investigational Site 15688, Hawthorne, New York
  - Teva Investigational Site 15603, Horseheads, New York
  - Teva Investigational Site 15666, Hyde Park, New York
  - Teva Investigational Site 15675, New Windsor, New York
  - Teva Investigational Site 15618, Asheville, North Carolina
  - Teva Investigational Site 15601, Chapel Hill, North Carolina
  - Teva Investigational Site 15697, Charlotte, North Carolina
  - Teva Investigational Site 15610, Elizabeth City, North Carolina
  - Teva Investigational Site 15651, High Point, North Carolina
  - Teva Investigational Site 15771, Statesville, North Carolina
  - Teva Investigational Site 15631, Wilmington, North Carolina
  - Teva Investigational Site 15584, Winston-Salem, North Carolina
  - Teva Investigational Site 15607, Cincinnati, Ohio
  - Teva Investigational Site 15613, Columbus, Ohio
  - Teva Investigational Site 15784, Dayton, Ohio
  - Teva Investigational Site 15791, Dayton, Ohio
  - Teva Investigational Site 15780, Toledo, Ohio
  - Teva Investigational Site 15662, Toledo, Ohio
  - Teva Investigational Site 15577, Oklahoma City, Oklahoma
  - Teva Investigational Site 15594, Tulsa, Oklahoma
  - Teva Investigational Site 15775, Yukon, Oklahoma
  - Teva Investigational Site 15646, Grants Pass, Oregon
  - Teva Investigational Site 15642, Philadelphia, Pennsylvania
  - Teva Investigational Site 15576, Pittsburgh, Pennsylvania
  - Teva Investigational Site 15608, North Charleston, South Carolina
  - Teva Investigational Site 15672, Rock Hill, South Carolina
  - Teva Investigational Site 15691, Knoxville, Tennessee
  - Teva Investigational Site 15705, Austin, Texas
  - Teva Investigational Site 15641, Boerne, Texas
  - Teva Investigational Site 15778, Brownsville, Texas
  - Teva Investigational Site 15668, Corsicana, Texas
  - Teva Investigational Site 15658, Dallas, Texas
  - Teva Investigational Site 15637, Dallas, Texas
  - Teva Investigational Site 15623, Dallas, Texas
  - Teva Investigational Site 15785, Edinburg, Texas
  - Teva Investigational Site 15678, El Paso, Texas
  - Teva Investigational Site 15787, El Paso, Texas
  - Teva Investigational Site 15591, El Paso, Texas
  - Teva Investigational Site 15696, Houston, Texas
  - Teva Investigational Site 15714, Houston, Texas
  - Teva Investigational Site 15680, Houston, Texas
  - Teva Investigational Site 15614, Houston, Texas
  - Teva Investigational Site 15578, Houston, Texas
  - Teva Investigational Site 15690, Katy, Texas
  - Teva Investigational Site 15684, Kerrville, Texas
  - Teva Investigational Site 15630, McKinney, Texas
  - Teva Investigational Site 15656, San Antonio, Texas
  - Teva Investigational Site 15670, San Antonio, Texas
  - Teva Investigational Site 15638, San Antonio, Texas
  - Teva Investigational Site 15647, Sherman, Texas
  - Teva Investigational Site 15673, Splendora, Texas
  - Teva Investigational Site 15707, Tomball, Texas
  - Teva Investigational Site 15693, Victoria, Texas
  - Teva Investigational Site 15649, Waxahachie, Texas
  - Teva Investigational Site 15671, Bountiful, Utah
  - Teva Investigational Site 15635, Sandy City, Utah
  - Teva Investigational Site 15789, West Valley City, Utah
  - Teva Investigational Site 15683, Williamsburg, Virginia
  - Teva Investigational Site 15586, Greenfield, Wisconsin
- Argentina (35):
  - Teva Investigational Site 20126, Bahía Blanca
  - Teva Investigational Site 20130, Bahía Blanca
  - Teva Investigational Site 20109, Bahía Blanca
  - Teva Investigational Site 20113, Buenos Aires
  - Teva Investigational Site 20135, Buenos Aires
  - Teva Investigational Site 20111, Buenos Aires
  - Teva Investigational Site 20138, Buenos Aires
  - Teva Investigational Site 20117, Buenos Aires Province
  - Teva Investigational Site 20128, CABA
  - Teva Investigational Site 20139, CABA
  - Teva Investigational Site 20129, CapitalFederal
  - Teva Investigational Site 20118, Concepción del Uruguay
  - Teva Investigational Site 20106, Córdoba
  - Teva Investigational Site 20125, Florida, Vicente Lopez
  - Teva Investigational Site 20136, Godoy Cruz
  - Teva Investigational Site 20122, Lanús Este
  - Teva Investigational Site 20107, Lobos
  - Teva Investigational Site 20123, Mar del Plata
  - Teva Investigational Site 20121, Mendoza
  - Teva Investigational Site 20115, Mendoza
  - Teva Investigational Site 20110, Mendoza
  - Teva Investigational Site 20127, Mendoza
  - Teva Investigational Site 20140, Paraná
  - Teva Investigational Site 20112, Quilmes
  - Teva Investigational Site 20119, Rosario
  - Teva Investigational Site 20105, Rosario
  - Teva Investigational Site 20120, Rosario
  - Teva Investigational Site 20133, San Fernando
  - Teva Investigational Site 20114, San Juan Bautista
  - Teva Investigational Site 20104, San Miguel de Tucumán
  - Teva Investigational Site 20124, San Miguel de Tucumán
  - Teva Investigational Site 20131, San Miguel de Tucumán
  - Teva Investigational Site 20137, San Miguel de Tucumán
  - Teva Investigational Site 20116, San Rafael
  - Teva Investigational Site 20132, Santa Fe
- Australia (8):
  - Teva Investigational Site 78131, Box Hill
  - Teva Investigational Site 78135, Clayton
  - Teva Investigational Site 78133, Melbourne
  - Teva Investigational Site 78132, Midland
  - Teva Investigational Site 78130, Nedlands
  - Teva Investigational Site 78134, North Adelaide
  - Teva Investigational Site 78128, Parkville
  - Teva Investigational Site 78127, South Brisbane
- Bulgaria (17):
  - Teva Investigational Site 59230, Blagoevgrad
  - Teva Investigational Site 59227, Kozloduy
  - Teva Investigational Site 59218, Pernik
  - Teva Investigational Site 59237, Pleven
  - Teva Investigational Site 59222, Plovdiv
  - Teva Investigational Site 59233, Plovdiv
  - Teva Investigational Site 59219, Rousse
  - Teva Investigational Site 59231, Sliven
  - Teva Investigational Site 59224, Sofia
  - Teva Investigational Site 59226, Sofia
  - Teva Investigational Site 59235, Sofia
  - Teva Investigational Site 59228, Sofia
  - Teva Investigational Site 59234, Sofia
  - Teva Investigational Site 59221, Sofia
  - Teva Investigational Site 59220, Stara Zagora
  - Teva Investigational Site 59232, Varna
  - Teva Investigational Site 59229, Vratsa
- Canada (6):
  - Teva Investigational Site 11267, Edmonton, Alberta
  - Teva Investigational Site 11272, Ajax, Ontario
  - Teva Investigational Site 11270, Etobicoke, Ontario
  - Teva Investigational Site 11274, Hamilton, Ontario
  - Teva Investigational Site 11271, Winchester, Ontario
  - Teva Investigational Site 11273, Windsor, Ontario
- Czechia (8):
  - Teva Investigational Site 54231, Brandýs nad Labem-Stará Boleslav
  - Teva Investigational Site 54232, Brno
  - Teva Investigational Site 54229, Jihlava
  - Teva Investigational Site 54226, Jindřichův Hradec
  - Teva Investigational Site 54225, Lovosice
  - Teva Investigational Site 54228, Ostrava
  - Teva Investigational Site 54230, Prague
  - Teva Investigational Site 54227, Varnsdorf
- Denmark (3):
  - Teva Investigational Site 39099, Aalborg
  - Teva Investigational Site 39100, Hvidovre
  - Teva Investigational Site 39098, Vejle
- Germany (26):
  - Teva Investigational Site 32846, Augsburg
  - Teva Investigational Site 32835, Berlin
  - Teva Investigational Site 32834, Berlin
  - Teva Investigational Site 32833, Berlin
  - Teva Investigational Site 32840, Cottbus
  - Teva Investigational Site 32829, Darmstadt
  - Teva Investigational Site 32850, Delitzsch
  - Teva Investigational Site 32853, Essen
  - Teva Investigational Site 32831, Frankfurt
  - Teva Investigational Site 32845, Frankfurt am Main
  - Teva Investigational Site 32838, Hamburg
  - Teva Investigational Site 32827, Hamburg
  - Teva Investigational Site 32848, Hamburg
  - Teva Investigational Site 32841, Hanover
  - Teva Investigational Site 32842, Heidelberg
  - Teva Investigational Site 32851, Ibbenbueren
  - Teva Investigational Site 32844, Leipzig
  - Teva Investigational Site 32830, Leipzig - Nordost
  - Teva Investigational Site 32832, Mainz A. Rhein
  - Teva Investigational Site 32847, München
  - Teva Investigational Site 32828, München
  - Teva Investigational Site 32843, Neu-Isenburg
  - Teva Investigational Site 32839, Neuss
  - Teva Investigational Site 32836, Peine
  - Teva Investigational Site 32849, Wiesbaden
  - Teva Investigational Site 32852, Witten
- Greece (7):
  - Teva Investigational Site 63086, Athens
  - Teva Investigational Site 63085, Evros
  - Teva Investigational Site 63089, Heraklion
  - Teva Investigational Site 63087, Larissa
  - Teva Investigational Site 63082, Thessaloniki
  - Teva Investigational Site 63083, Thessaloniki
  - Teva Investigational Site 63088, Thivon and Livadias
- Hungary (8):
  - Teva Investigational Site 51346, Budapest
  - Teva Investigational Site 51344, Budapest
  - Teva Investigational Site 51340, Budapest
  - Teva Investigational Site 51342, Debrecen
  - Teva Investigational Site 51345, Mosonmagyaróvár
  - Teva Investigational Site 51343, Pécs
  - Teva Investigational Site 51339, Szeged
  - Teva Investigational Site 51341, Szigetvár
- Israel (9):
  - Teva Investigational Site 80196, Ashkelon
  - Teva Investigational Site 80201, Beersheba
  - Teva Investigational Site 80200, Haifa
  - Teva Investigational Site 80194, Jerusalem
  - Teva Investigational Site 80198, Jerusalem
  - Teva Investigational Site 80199, Petach Tikvah
  - Teva Investigational Site 80195, Petah Tikva
  - Teva Investigational Site 80193, Rehovot
  - Teva Investigational Site 80197, Tel Aviv
- Italy (5):
  - Teva Investigational Site 30306, Ferrara
  - Teva Investigational Site 30316, Padua
  - Teva Investigational Site 30317, Pisa
  - Teva Investigational Site 30318, Verona
  - Teva Investigational Site 30307, Verona
- Latvia (8):
  - Teva Investigational Site 56016, Balvi
  - Teva Investigational Site 56019, Daugavpils
  - Teva Investigational Site 56017, Jūrmala
  - Teva Investigational Site 56015, Rēzekne
  - Teva Investigational Site 56014, Riga
  - Teva Investigational Site 56013, Riga
  - Teva Investigational Site 56020, Riga
  - Teva Investigational Site 56018, Riga
- Mexico (6):
  - Teva Investigational Site 21125, Chihuahua City
  - Teva Investigational Site 21122, Guadalajara
  - Teva Investigational Site 21127, Guadalajara
  - Teva Investigational Site 21126, Monterrey
  - Teva Investigational Site 21123, Oaxaca City
  - Teva Investigational Site 21129, Villahermosa
- New Zealand (12):
  - Teva Investigational Site 79054, Auckland
  - Teva Investigational Site 79056, Auckland
  - Teva Investigational Site 79055, Christchurch
  - Teva Investigational Site 79057, Dunedin
  - Teva Investigational Site 79051, Hamilton
  - Teva Investigational Site 79062, Nawton
  - Teva Investigational Site 79061, Nelson
  - Teva Investigational Site 79059, Rotorua
  - Teva Investigational Site 79060, South Hastings
  - Teva Investigational Site 79052, Tauranga
  - Teva Investigational Site 79058, Waikanae Beach
  - Teva Investigational Site 79050, Wellington
- Poland (18):
  - Teva Investigational Site 53531, Bialystok
  - Teva Investigational Site 53527, Bialystok
  - Teva Investigational Site 53534, Bydgoszcz
  - Teva Investigational Site 53537, Elblag
  - Teva Investigational Site 53524, Gdansk
  - Teva Investigational Site 53538, Gdansk
  - Teva Investigational Site 53530, Krakow
  - Teva Investigational Site 53521, Krakow
  - Teva Investigational Site 53528, Lodz
  - Teva Investigational Site 53523, Lublin
  - Teva Investigational Site 53533, Lublin
  - Teva Investigational Site 53522, Maków Podhalański
  - Teva Investigational Site 53525, Ostrowiec Świętokrzyski
  - Teva Investigational Site 53532, Poznan
  - Teva Investigational Site 53526, Rzeszów
  - Teva Investigational Site 53536, Skierniewice
  - Teva Investigational Site 53535, Warsaw
  - Teva Investigational Site 53529, Zawadzkie
- Romania (6):
  - Teva Investigational Site 52139, Bacau
  - Teva Investigational Site 52140, Bragadiru
  - Teva Investigational Site 52138, Bucharest
  - Teva Investigational Site 52136, Bucharest
  - Teva Investigational Site 52135, Cluj-Napoca
  - Teva Investigational Site 52137, Craiova
- Serbia (11):
  - Teva Investigational Site 61071, Belgrade
  - Teva Investigational Site 61073, Belgrade
  - Teva Investigational Site 61074, Belgrade
  - Teva Investigational Site 61075, Belgrade
  - Teva Investigational Site 61080, Belgrade
  - Teva Investigational Site 61076, Belgrade
  - Teva Investigational Site 61077, Belgrade
  - Teva Investigational Site 61072, Kamenitz
  - Teva Investigational Site 61078, Kragujevac
  - Teva Investigational Site 61070, Niš
  - Teva Investigational Site 61079, Novi Sad
- Slovakia (7):
  - Teva Investigational Site 62083, Bardejov
  - Teva Investigational Site 62082, Košice
  - Teva Investigational Site 62080, Rimavská Sobota
  - Teva Investigational Site 62077, Slovakia
  - Teva Investigational Site 62078, Spišská Nová Ves
  - Teva Investigational Site 62079, Žilina
  - Teva Investigational Site 62081, Žilina
- South Africa (21):
  - Teva Investigational Site 90078, Benoni
  - Teva Investigational Site 90069, Cape Town
  - Teva Investigational Site 90077, Cape Town
  - Teva Investigational Site 90063, Cape Town
  - Teva Investigational Site 90079, Cape Town
  - Teva Investigational Site 90073, Chatsworth
  - Teva Investigational Site 90067, Durban
  - Teva Investigational Site 90070, Ennerdale
  - Teva Investigational Site 90083, Germiston
  - Teva Investigational Site 90062, Johannesburg
  - Teva Investigational Site 90074, Krugersdorp
  - Teva Investigational Site 90065, KwaDukuza
  - Teva Investigational Site 90064, Middelburg
  - Teva Investigational Site 90072, Midrand
  - Teva Investigational Site 90071, Plettenberg Bay
  - Teva Investigational Site 90081, Polokwane
  - Teva Investigational Site 90076, Pretoria
  - Teva Investigational Site 90080, Raslouw
  - Teva Investigational Site 90068, Roodepoort
  - Teva Investigational Site 90066, Somerset West
  - Teva Investigational Site 90082, Soweto
- South Korea (6):
  - Teva Investigational Site 87039, Seoul
  - Teva Investigational Site 87044, Seoul
  - Teva Investigational Site 87043, Seoul
  - Teva Investigational Site 87042, Seoul
  - Teva Investigational Site 87040, Seoul
  - Teva Investigational Site 87041, Seoul
- Spain (9):
  - Teva Investigational Site 31304, Badalona
  - Teva Investigational Site 31305, Barcelona
  - Teva Investigational Site 31307, Barcelona
  - Teva Investigational Site 31309, Córdoba
  - Teva Investigational Site 31303, Madrid
  - Teva Investigational Site 31310, Sabadell
  - Teva Investigational Site 31306, Santiago de Compostela
  - Teva Investigational Site 31311, Seville
  - Teva Investigational Site 31308, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.